CLINICAL TRIAL: NCT05848518
Title: Effect of Different Types of Supervised Exercise Programs on Cardiorespiratory and Muscular Fitness, Pain, Fatigue, Mental Health and Inflammatory and Oxidative Stress Biomarkers in Older COVID-19 Survivors. (EJerSA-COVID-19)
Brief Title: Exercise for Health in Patients With Post-acute Sequelae of COVID-19
Acronym: EJerSA-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus docent Sant Joan de Déu-Universitat de Barcelona (Other)
Collaborators: Hospital de Mataró (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Manuel Vicente Garnacho Castano, Coordinator of the DAFNiS research group, Campus docent Sant Joan de Déu-Universitat de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CampusSantJoan
Record Dates: First submitted 2023-05-02; First posted 2023-05-08 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Long COVID
Keywords: rehabilitation programs; endurance exercise; resistance exercise; cardiopulmonary exercise testing; muscle strength assessment; quality of life; elderly people; severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Concurrent rehabilitation program (Experimental): Endurance plus resistance exercises
  Interventions: Other: Rehabilitation program
- Endurance rehabilitation program (Experimental): Endurance exercises
  Interventions: Other: Rehabilitation program
- Strength rehabilitation program (Experimental): Resistance exercises
  Interventions: Other: Rehabilitation program
- Control group (No Intervention): No exercise

INTERVENTIONS:
Other: Rehabilitation program — The participants will be randomly assigned to the experimental groups: supervised endurance rehabilitation program (SEG, n = 30), supervised strength rehabilitation program (SSG, n = 30), supervised concurrent rehabilitation program (SCG, n = 30), and control group (CG, n = 30)
  Arms: Concurrent rehabilitation program; Endurance rehabilitation program; Strength rehabilitation program

SUMMARY:
Background: Many patients with COVID-19 present the so-called post-acute sequelae of COVID-19 such as fatigue, post-stress discomfort, dyspnea, headache, pain mental impairment, incapacity to perform daily physical tasks ant exercise intolerance. This study aims to investigate the effects of different exercise programs on physical and mental fitness, physical condition and biomarkers of the immune system and oxidative stress in older COVID-19 survivors. Methods: The sample will be made up of 120 eligible participants, over the age of 60 years who have had COVID-19 disease and are survivors and present persistent COVID-19 symptomatology diagnosed by the corresponding physician. The participants will be randomly assigned to the experimental groups: supervised endurance group (SEG, n = 30), supervised strength group (SSG, n = 30), supervised concurrent group (SCG, n = 30), which will perform the corresponding exercise program 3 days a week compared to the control group (CG, n = 30), which will not carry out a supervised exercise program. The design of this project will include assessment of cardiorespiratory fitness, muscle fitness, pain and mental health, and biomarkers of inflammation and oxidative stress.

DETAILED DESCRIPTION:
This project will carry out a randomized controlled trial to determine what type of supervised exercise program is the most effective compared with a control group (CG): supervised endurance group (SEG), supervised strength group (SSG), supervised concurrent group (strength and endurance) (SCG) and CG. The project will be divided into 3 subprojects and performed in coordination by three institutions as follows:

i) Subproject of the consolidated research group on pain, physical activity, nutrition and health (Acronym: DAFNiS) of the Campus Sant Joan de Deu. University of Barcelona. "Effects of a physical exercise program (aerobic, strength or combined/concurrent) on muscle fitness, pain and mental health in older COVID-19 survivors".

ii) Subproject of the Hospital of Matar: "Evaluation of cardiorespiratory and muscular fitness in older COVID-19 survivors".

iii) Subproject of the Department of Physiology and Immunology. University of Barcelona. "Evaluation of biomarkers of inflammation and oxidative stress in older COVID-19 survivors".

The sample will be made up of 120 eligible participants, over the age of 60 years who have had COVID-19 disease and are survivors and present persistent COVID-19 symptomatology with sequelae of fatigue, muscle weakness, pain, difficulty in performing daily life activities, etc. diagnosed by the corresponding physician. The participants will be recruited from Hospital of Matar. Candidates fulfilling the study inclusion criteria will provide signed informed consent prior to inclusion.

To calculate the sample size of this project a type 1 (α) error of 5% and a 95% confidence interval with a level of precision (d = 0.095) was established for the test of proportional hypotheses resulting in a sample size of n= 108 persons, increased by 10% (rounded up to n=120) to compensate for possible dropouts along the study period.

To know the sample size more precisely in the hypothesis test of means it will be necessary to carry out a pilot study which will provide the size of effect and statistical power (0.80), determine the analysis to perform, obtain delta values in the units corresponding to the principal study variable as well as know the standard deviation.

Program of supervised exercise The intervention will consist in a program of supervised physical exercise performed 3 times a week for 12 weeks. For the planning and control of the exercise program the progressive individualized planning model will be applied based on the subjective perception of effort and cardiorespiratory parameters (heart rate and ventilatory threshold determined in the evaluation tests) of the participants. This program has been used by our research group in previous studies for improving cardiorespiratory and muscle fitness. The basis of this periodization model establishes an initial period of individualization to obtain the personal parameters used for the training load

The COVID-19 survivors will be randomly assigned to 3 programs of supervised exercise :

1. Program of endurance exercise. The program of supervised endurance exercise will consist in walking for 1 hour 3 times a week. The intensity (step speed) will gradually be increased each week (approx. 5%) according to the perception of the participant. A pulsometer will be used to determine the safe range of heart rate at which the participant should perform.
2. Program of strength exercise This will consist in performing a program of traditional strength 1 hour 3 times a week. Circuit training methodology will be used (10 exercises) alternating muscle groups of the upper and lower extremities and trunk. The initial series be of 1 exercise, evolving to up to 3-4 along the program based on the individual adaptation of the individual. The intensity (load applied) will be gradually increased each week while the recovery times between each exercise activity will be reduced (approx. 5%) according to the perception of the participant. A pulsometer will be used to determine the safe range of heart rate at which the participant should perform.
3. Program of concurrent exercise (endurance and strength) The participants will perform 1 hour of concurrent exercise, combining walking (20 minutes) and the strength program for 40 minutes, maintaining the same instructions explained previously in each exercise program.
4. Control group The control group will not carry out any supervised exercise program but will maintain their same habits of daily life activities.

Process of evaluation To determine the effects of the exercise program, an initial evaluation will be made before beginning the exercise program to assess the initial status of the participants (Pre). This evaluation will be compared with the evaluation made at the end of the intervention program (Post) at 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Persons of both sexes (and different expression of gender) older than 60 years of age.
* No history of physical diseases and no disease or disability that limits participation in the exercise program or precludes the corresponding measurement/evaluations.
* Be able to communicate without difficulty.
* Be able to understand the objectives of the project and provide informed consent. In this case, the consent form will be signed.
* Not taking any medication that can affect normal performance of the exercise program and the evaluations

Exclusion Criteria:

* Having acute or terminal disease or any other disease that may affect the normal practice of a supervised exercise program and the corresponding evaluations.
* Consumption of alcohol or drugs.
* Be performing any type of activity that may interfere in carrying out the supervised exercise program or the evaluations.
* Not completing the study once initiated or wishing to participate in the control group.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness: absolute oxygen uptake | 1 week per group
  absolute oxygen uptake (peak VO2) in L/min
Cardiorespiratory fitness: relative oxygen uptake | 1 week per group
  relative oxygen uptake (peak VO2) in mL/kg/min
Cardiorespiratory fitness: ventilation | 1 week per group
  minute ventilation (VE) in L/min.
Cardiorespiratory fitness: ventilatory equivalent for oxygen | 1 week per group
  Ventilatory equivalent for oxygen (VE/VO2)
Cardiorespiratory fitness: ventilatory equivalent for carbon dioxide | 1 week per group
  Ventilatory equivalent for carbon dioxide (VE/VCO2)
Cardiorespiratory fitness: respiratory exchange ratio | 1 week per group
  Respiratory exchange ratio (RER)
Cardiorespiratory fitness: End-tidal partial pressure | 1 week per group
  End-tidal partial pressure of oxygen and carbon dioxide (PetO2 and PetCO2, respectively) in mmHg.
Muscular fitness: Sit and stand test | 1 week per group
  Sit and stand test for 30 seconds. The number of times in 30 seconds the participant can completely stand up from a seated position with the back straight and the feet on the floor without pushing with the arms will be counted.
Muscular fitness: countermovement jump | 1 week per group
  Countermovement jumps: Flight Height in cm
Muscular fitness: countermovement test | 1 week per group
  Countermovement jumps: power output of the lower extremities in watts
Muscular fitness: Upper limb strength | 1 week per group
  This will be evaluated with the bicep curl test made with a 2 kg weight for women and a 4 Kg weight for men. The number of elbow curls made in 30 seconds with each upper limb will be counted.
Muscular fitness: hand grip strength | 1 week per group
  Hand grip strength: Force in Newtons Motor Agility/Dynamic balance: This will be evaluated with the 8-foot up and go test. The best of two attempts will be registered
Muscular fitness: Motor Agility/Dynamic balance | 1 week per group
  Motor Agility/Dynamic balance: This will be evaluated with the 8-foot up and go test. The best of two attempts will be registered in seconds
Muscular fitness: Isokinetic strength test | 1 week per group
  The isokinetic knee flexor and extensor test: peak torque in N m
Muscular fitness: Isokinetic strength testing | 1 week per group
  The isokinetic knee flexor and extensor test: power output in Watts
Body composition: fat mass | 1 week per group
  Fat mass will be assessed by bioelectrical impedance analysis in kg and percentage of body weight.
Body composition: fat free mass | 1 week per group
  Fat free mass will be assessed by bioelectrical impedance analysis in kg and percentage of body weight.
Body composition: muscle mass | 1 week per group
  Muscle mass will be assessed by bioelectrical impedance analysis in kg and percentage of body weight.
Concentration of oxidative stress biomarkers: thiobarbituric acid reactive substances | 1 week per group
  Determination of oxidized lipids by the thiobarbituric acid reactive substances (TBARS) in mmols (fluorimetry technique).
Concentration of oxidative stress biomarkers: Advanced Oxidation Protein Products | 1 week per group
  Determination of oxidized proteins by the Advanced Oxidation Protein Products (AOPP) in nmol Cl-T/mg protein, (colorimetry technique)
Concentration of oxidative stress biomarkers: nitrites and nitrates | 1 week per group
  Determination of nitrites and nitrates (colorimetry) in nmol/mL
Concentration of biomarkers of antioxidant enzymes: superoxide dismutase | 1 week per group
  superoxide dismutase (SOD) in units/mL
Concentration of biomarkers of antioxidant enzymes: catalase | 1 week per group
  catalase (CAT) in units/mL
Concentration of biomarkers of antioxidant enzymes: glutathion peroxidase | 1 week per group
  Glutathion peroxidase (GPx) in units/mL.
Concentration of inflammation biomarkers: Interleukines | 1 week per group
  Interleukin 6 and 10 (IL-6 and IL-10) in ng/mL
Concentration of inflammation biomarkers: adiponectin | 1 week per group
  adiponectin in mg/L
Concentration of biomarkers of inflammation: Tumor necrosis factor | 1 week per group
  Tumor Necrosis Factor-alpha in pg/mL
Evaluation of the degree of pain using the pupillometer: pupil diameter | 1 week per group
  basal and maximum diameter of the pupil in mm
Evaluation of the degree of pain using the pupillometer:variation of pupil | 1 week per group
  percentage of variation of pupil diameter in %
Evaluation of the degree of pain using the pupillometer: pupil variation | 1 week per group
  variation of the pupil in mm
Evaluation of the degree of pain using the pupillometer: Intensity of reflex of dilatation | 1 week per group
  Intensity of reflex of dilatation, latency.
Evaluation of the degree of pain with a pressure algometer: algometers | 1 week per group
  Pain will be quantified with a pressure algometer + pupillometer in older COVID-19 survivors.
  A pressure algometer allows the application of a controlled and quantifiable nociceptive stimulus on a body surface.
  Algometers apply a pressure stimulus that can be useful for applying a standardized painful stimulus, having a different nature from that applied with the pupillometer which is a stimulus of electric origin.
Mental health | 1 week per group
  Psychosocial variables will be evaluated using the Hospital Anxiety and Depression Scale (HADS), which is made up of 7 items for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) will be scored on a scale of 4 points from 0 (none) to 3 (much more). The highest scores indicate the highest levels of anxiety or depression

CONTACTS AND LOCATIONS:
Overall Officials: Manuel V Garnacho-Castaño, PhD, Principal Investigator — Campus docent Sant Joan de Déu-Universitat de Barcelona
Locations (1):
- Campus Docent Sant Joan de Déu. Universitat de Barcelona, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pleguezuelos E, Sanchez-Nuno S, Del Carmen A, Serra-Paya N, Moreno E, Molina-Raya L, Robleda G, Benet M, Santos-Ruiz S, Garrido AB, Jerez-Molina C, Miravitlles M, Serra-Prat M, Vinals X, Farres MG, Carbonell T, Garnacho-Castano MV. Effect of different types of supervised exercise programs on cardiorespiratory and muscular fitness, pain, fatigue, mental health and inflammatory and oxidative stress biomarkers in older patients with post-COVID-19 sequelae "EJerSA-COVID-19": a randomized controlled trial. BMC Geriatr. 2023 Dec 15;23(1):865. doi: 10.1186/s12877-023-04544-3. PMID 38102536